CLINICAL TRIAL: NCT00697788
Title: Cardiovascular Safety of Dexmedetomidine in Pediatric Burn Patients.
Brief Title: Dexmedetomidine Cardiovascular Safety in Pediatric Burn Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Erik S. Shank, MD, Pediatric Anesthesiologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-P-001264/1;MGH
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-06

CONDITIONS: Burns; Sedation
Keywords: pediatric; burn; sedation
MeSH Terms: conditions — Burns | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ascending dose study (Experimental): Ascending doses of dexmedetomidine (as per protocol)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine bolus 1 ug/kg over 10 minutes, followed by ascending infusion as follows: Dexmedetomidine [in ug/kg/hr], each for 15 minutes: 0.7, 1.0, 1.3, 1.6, 1.9, 2.2, 2.5.
  Other Names: Precedex

SUMMARY:
Dexmedetomidine is a sedative drug approved for adult patients, intubated, in intensive care units. We are studying whether this drug is cardiovascularly safe in pediatric patients who have recently been burned.

DETAILED DESCRIPTION:
This is an ascending dose study evaluating the cardiovascular safety of dexmedetomidine bolus/infusions in acutely burned pediatric patients. The study entails a bolus of dexmedetomidine, followed by 2 hours of increasing infusion doses. Cardiovascular parameters including EKG, heart rate, oxygen saturation, blood pressure, are recorded.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patient
* >25% total body surface area (tbsa) burn and < 90% tbsa
* opioid requirements > 0.1 mg/kg/hour of morphine (or equivalent)
* midazolam requirement > 0.1 mg/kg/hour
* treatment team determined that patient should be started on dexmedetomidine

Exclusion Criteria:

* hemodynamically unstable patients (epinephrine > 1.0 ug/kg/min, levophed > 0.75 ug/kg/min, dopamine > 10 ug/kg/min)
* pregnant patients
* patients with history of heart block
* patients with congenital heart disease
* patients with significant hepatic dysfunction
* patients with urine output < 0.5 ml/kg/hour [averaged] over past 24 hours

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2007-07-16 (Actual); Primary Completion 2008-12-30 (Actual); Study Completion 2008-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik S Shank, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Shriners Burn Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV: All participants received a dexmedetomidine bolus of 1.0 micrograms (mcg) per kilogram over 10 minutes.
- Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion: This group received the bolus dose and a continuous infusion for 15 minutes of 0.7 mcg/kg/hr of dexmedetomidine. This group is a subset of Cohort 1 that continued in this ascending dose study.
- Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion: This group received the bolus dose, followed by dexmedetomidine infusion for 15 minutes at 0.7 mcg/kg/hr, followed by 1.0 mcg/kg/hr infusion for 15 minutes. This is a subset of cohort 2.
- Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr: This group received the bolus dose followed by the ascending infusion first at 0.7 mcg/kg/hr for 15 minutes, then 1.0 mcg/kg/hr for 15 minutes, the 1.3 mcg/kg.hr for 15 minutes. This group is a subset of cohort 3.
- Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion: This group received the bolus dose followed by the ascending infusion first at 0.7 mcg/kg/hr for 15 minutes, then 1.0 mcg/kg/hr for 15 minutes, the 1.3 mcg/kg.hr for 15 minutes, followed by 1.6 mcg/kg/hr for 15 minutes. This group is a subset of cohort 4.
- Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr: This group received the bolus dose followed by the ascending infusion first at 0.7 mcg/kg/hr for 15 minutes, then 1.0 mcg/kg/hr for 15 minutes, the 1.3 mcg/kg.hr for 15 minutes, followed by 1.6 mcg/kg/hr for 15 minutes, followed by 1.9 mcg/kg/hr for 15 minutes. This group is a subset of cohort 5.
- Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr: This group received the bolus dose followed by the ascending infusion first at 0.7 mcg/kg/hr for 15 minutes, then 1.0 mcg/kg/hr for 15 minutes, the 1.3 mcg/kg.hr for 15 minutes, followed by 1.6 mcg/kg/hr for 15 minutes, followed by 1.9 mcg/kg/hr for 15 minutes, followed by 2.2 mcg/kg/hr over 15 minutes. This group is a subset of cohort 6.
- Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr: This group received the bolus dose followed by the ascending infusion first at 0.7 mcg/kg/hr for 15 minutes, then 1.0 mcg/kg/hr for 15 minutes, the 1.3 mcg/kg.hr for 15 minutes, followed by 1.6 mcg/kg/hr for 15 minutes, followed by 1.9 mcg/kg/hr for 15 minutes, followed by 2.2 mcg/kg/hr over 15 minutes, followed by 2.5 mcg/kg/hr over 15 minutes. This group is a subset of cohort 7.
Period: Dexmedetomidine Bolus 1 mcg/kg
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Started | 8 | 0 (One participant did not begin infusion due to hypotension (mean pressure <50)) | 0 (2 participants did not begin the ascending (1.0 mcg/kg/hr) due to MAP<50) | 0 | 0 | 0 | 0 | 0
Completed | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dexmedetomidine 0.7 mcg/kg/hr Infusion
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Started | 0 | 7 (1 participant did not begin infusion due to hypotension (MAP<50)) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dexmedetomidine 1.0 mcg/kg/hr Infusion
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Started | 0 | 0 | 3 (2 participants did not begin this infusion due to hypotension (MAP<50)) | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dexmedetomidine 1.3 mcg.kg/hr Infusion
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Started | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dexmedetomidine 1.6 mcg.kg.hr Infusion
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Started | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Dexmedetomidine 1.9 mcg/kg/hr Infusion
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Started | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dexmedetomidine 2.2 mcg/kg/hr Infusion
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Started | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dexmedetomidine 2.5 mcg/kg/hr Infusion
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ascending Dose Study
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Total Body Surface Area Burned [Mean (Standard Deviation); unit: percentage of surface] | 58.3 (15.2)
Weight [Mean (Standard Deviation); unit: kilograms] | 33.5 (23.5)
Central Venous Pressure [Mean (Standard Deviation); unit: millimeters of mercury (mm Hg)] | 10.4 (4)
Time after injury in days [Mean (Standard Deviation); unit: days] | 19.7 (10.3)
Fluid intake-Fluid output [Mean (Standard Deviation); unit: ml/kg/24 hours] | 88.7 (71.8)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Mean Arterial Pressure (MAP)
Description: Looking at hemodynamic response to dexmedetomidine. Mean arterial pressure primary outcome measure.
Time Frame: 10, 25, 40, 55, 70, 85, 100, 115 minutes after dexmedetomidine bolus administration
Population: Acutely burned pediatric patients intubated with burns >=20% between 2 and 19 years of age requiring escalating doses of morphine and midazolam
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine Bolus + 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Number analyzed (Participants) | 8 | 5 | 4 | 4 | 4 | 3 | 3 | 3
% change | 26.7 (7.5) | 30.8 (10.2) | 26.5 (10.5) | 24.5 (13.8) | 25.5 (12.5) | 18 (8.7) | 15 (7) | 15.6 (8.0)

2. Secondary Outcome: Presence of Arrhythmias.
Description: Presence of arrhythmias was studied using a 3 lead realtime EKG throughout study.
Time Frame: 10, 25, 40, 55, 70, 85, 100, 115 minutes after dexmedetomidine bolus administration
Population: EKG was analyzed on each participant looking for presence of arrhythmias. None were detected.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV: Ascending doses of dexmedetomidine (as per protocol)
  Dexmedetomidine: Dexmedetomidine bolus 1 ug/kg over 10 minutes, followed by ascending infusion as follows: Dexmedetomidine [in ug/kg/hr], each for 15 minutes: 0.7, 1.0, 1.3, 1.6, 1.9, 2.2, 2.5.
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine Bolus + 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Number analyzed (Participants) | 8 | 5 | 4 | 4 | 4 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Oxygen Saturation
Description: Pulse oximetry was used to measure oxygen saturation.
Time Frame: 10, 25, 40, 55, 70, 85, 100, 115 minutes after dexmedetomidine bolus administration
Measure: Mean (Standard Deviation); unit: Percent of Hemoglobin Saturated
Groups:
- Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion: This group received the bolus dexmedetomidine and a continuous infusion for 15 minutes of 0.7 mcg/kg/hr of dexmedetomidine. This group is a subset of Cohort 1 that continued in this ascending dose study.
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Number analyzed (Participants) | 8 | 5 | 4 | 4 | 4 | 3 | 3 | 3
Percent of Hemoglobin Saturated | 99.8 (0.5) | 99.5 (0.8) | 99.5 (0.8) | 98.6 (1.1) | 98.6 (1.1) | 98.6 (1.3) | 99.3 (1.5) | 99.5 (0.6)

4. Secondary Outcome: Heart Rate
Description: Heart Rate recorded off EKG in beats per minute
Time Frame: 10, 25, 40, 55, 70, 85, 100, 115 minutes after dexmedetomidine bolus administration
Measure: Mean (Standard Deviation); unit: heart beats per minute
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine Infusion 1.3 mcg/kg/hr | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr
Number analyzed (Participants) | 8 | 5 | 4 | 4 | 4 | 3 | 3 | 3
heart beats per minute | 125.6 (16.6) | 122 (15.8) | 127.5 (11.9) | 125.5 (17.2) | 122.8 (17.8) | 129.7 (11.6) | 132.3 (17.9) | 125 (8.9)

ADVERSE EVENTS:
Time Frame: Data was collected for the two hour period of the study.
Groups:
- Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV: All participants received a dexmedetomidine bolus dose of 1 microgram/kilogram over 10 minutes IV
- Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion: This group received the bolus dose and then an infusion of 0.7 mcg/kg/hr for 15 minutes
- Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion: This group received the bolus dose and then an infusion of 0.7 mcg/kg/hr for 15 minutes, followed by 1.0 mcg/kg/hr over 15 minutes
- Cohort 4: Dexmedetomidine 1.3 mcg/kg/hr Infusion: This group received the bolus dose and then an infusion of 0.7 mcg/kg/hr for 15 minutes, followed by 1.0 mcg/kg/hr over 15 minutes, followed by 1.3 mcg/kg/hr
- Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion: This group received the bolus dose and then an infusion of 0.7 mcg/kg/hr for 15 minutes, followed by 1.0 mcg/kg/hr over 15 minutes, followed by 1.3 mcg/kg/hr, followed by 1.6 mcg/kg/hr over 15 minutes
- Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr Infusion: This group received the bolus dose and then an infusion of 0.7 mcg/kg/hr for 15 minutes, followed by 1.0 mcg/kg/hr over 15 minutes, followed by 1.3 mcg/kg/hr, followed by 1.6 mcg/kg/hr over 15 minutes, followed by 1.9 mcg/kg/hr over 15 minutes
- Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr Infusion: This group received the bolus dose and then an infusion of 0.7 mcg/kg/hr for 15 minutes, followed by 1.0 mcg/kg/hr over 15 minutes, followed by 1.3 mcg/kg/hr, followed by 1.6 mcg/kg/hr over 15 minutes, followed by 1.9 mcg/kg/hr over 15 minutes, followed by 2.2 mcg/kg/hr over 15 minutes
- Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr Infusion: This group received the bolus dose and then an infusion of 0.7 mcg/kg/hr for 15 minutes, followed by 1.0 mcg/kg/hr over 15 minutes, followed by 1.3 mcg/kg/hr, followed by 1.6 mcg/kg/hr over 15 minutes, followed by 1.9 mcg/kg/hr over 15 minutes, followed by 2.2 mcg/kg/hr over 15 minutes, followed by 2.5 mcg/kg/hr over 15 minutes
Arm/Group | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion | Cohort 4: Dexmedetomidine 1.3 mcg/kg/hr Infusion | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr Infusion | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr Infusion | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr Infusion
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/4 | 0/4 | 0/4 | 0/3 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/4 | 0/4 | 0/4 | 0/3 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/8 | 2/7 | 0/4 | 0/4 | 0/4 | 0/3 | 0/3 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Dexmedetomidine Bolus 1 mcg/kg Over 10 Min IV (N=8) | Cohort 2: Dexmedetomidine 0.7 mcg/kg/hr Infusion (N=7) | Cohort 3: Dexmedetomidine 1.0 mcg/kg/hr Infusion (N=4) | Cohort 4: Dexmedetomidine 1.3 mcg/kg/hr Infusion (N=4) | Cohort 5: Dexmedetomidine 1.6 mcg/kg/hr Infusion (N=4) | Cohort 6: Dexmedetomidine 1.9 mcg/kg/hr Infusion (N=3) | Cohort 7: Dexmedetomidine 2.2 mcg/kg/hr Infusion (N=3) | Cohort 8: Dexmedetomidine 2.5 mcg/kg/hr Infusion (N=2)
Significant hypotension defined as mean arterial pressure <50 mm Hg (Vascular disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 — Hypotension, defined as mean arterial pressure (MAP) < 50 millimeters of mercury, was considered an adverse event and would halt the ascending dose study for the subject.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes